CLINICAL TRIAL: NCT02346487
Title: Prospective Study of Lopinavir Based ART for HIV Infected childreN Globally
Brief Title: Prospective Study of Lopinavir Based ART for HIV Infected childreN Globally (LIVING Study)
Acronym: LIVING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: UNITAID (Other); French Development Agency (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNDiHIVPed002
Record Dates: First submitted 2015-01-13; First posted 2015-01-27 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: HIV
Keywords: children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LPV/RTV pellets and AZT/3TC or ABC/3TC (Experimental): Only 1 arm. No comparator
  Interventions: Drug: LPV/RTV pellets and AZT/3TC or ABC/3TC

INTERVENTIONS:
Drug: LPV/RTV pellets and AZT/3TC or ABC/3TC — Drug: LPV/r pellets 40/10 mg: orally taken twice a day. Dosage according to patient's weight:
  * Between 3 and 5.9kg: 2 capsules twice a day
  * Between 6 and 9.9kg: 3 capsules twice a day
  * Between 10 and 13.9kg: 4 capsules twice a day
  * Between 14 and 19.9kg: 5 capsules twice a day
  * Between 20 and 24.9kg: 6 capsules twice a day
  Drug: NRTIs (AZT/3TC 60/30mg tablet or ABC/3TC 60/30mg tablet). Dosage according to patient's weight:
  * Between 3 and 5.9kg: 1 tablet twice a day
  * Between 6 and 9.9kg: 1.5 tablets twice a day
  * Between 10 and 13.9kg: 2 tablets twice a day
  * Between 14 and 19.9kg: 2.5 tablets twice a day
  * Between 20 and 24.9kg: 3 tablets twice a day

SUMMARY:
The study will be carried out to provide supportive clinical data on the feasibility, efficacy, safety, and PK of LPV based therapies in routine treatment setting and will be based on the existing LPV/r pellets which already represent a clear advantage in comparison with the liquid formulation.

DETAILED DESCRIPTION:
The primary objective is to evaluate the effectiveness of LPV/r pellets in addition to AZT/3TC (or ABC/3TC) paediatric fixed dose combination (FDCs) tablet under routine treatment conditions in HIV infected infants and young children who cannot swallow tablets.

As secondary objectives:

* Document the safety of LPV/r pellets and AZT/3TC or ABC/3TC
* Assess the population pharmacokinetics of LPV/r and NRTIs when administered as LPV/r pellets plus AZT/3TC or ABC/3TC
* Measure adherence to the new formulation
* Evaluate children acceptability of the LPV/r pellets and associated dual NRTIs as well as ease of use by the care giver.

ELIGIBILITY:
Inclusion Criteria:

• Past or current documentation of a confirmed diagnosis of HIV infection defined as two positive assays from two different samples taken at a different date as preferred option.

* At any age: HIV-1 DNA PCR positivity
* At any time >4 weeks of age: HIV-1 p24 antigen detection or HIV-1 RNA viral load > 5,000 copies/mL plasma
* At any age >18 months: HIV-1 antibody reactive on two different manufacturers' licensed rapid tests based on a different antigen preparation and/or different test principal, or repeatedly reactive on a licensed enzyme immune assay (EIA)and confirmed on a second sample by any one of the following assays: rapid test (a third manufacturer), licensed EIA, Western blot, chemi-luminescence assay, or plasma RNA with a viral load > 5,000 copies/mL

One single positive PCR assay result will be acceptable for inclusion of a child less than 18 months in the study Although the 2nd PCR assay would not be performed at the time of treatment initiation/treatment switch,

* In case the test is RNA PCR viral load), the sample should be taken before treatment initiation and analyzed as soon as possible thereafter,
* In case the child is already on treatment, the test should be DNA PCR based, the blood sample can be taken while on treatment and the results be made available as soon as possible.
* ARV treatment eligible children with LPV-based treatment indication* as defined by country-specific guidelines or the WHO pediatric treatment guidelines confirmed by investigator:

  1. ARV naïve, or
  2. Already on first line liquid lopinavir based treatment, or
  3. Failing first line NNRTI based therapy
* Weight ≥3 and <25 kg at the time of enrolment.
* Inability to swallow tablets*
* Parent or legal guardian able and willing to provide written informed consent. *Age is not an inclusion criterion. Children older than 5 years who need a LPV/r based treatment and cannot swallow tablets are eligible. Analysis will be stratified according to study entry point (naïve, first line, failure)

Exclusion criteria

* Planned or concurrent use of NNRTIs, integrase inhibitors, entry inhibitors, or PIs other than LPV/r.
* PIs treatment failure with the presence or strong suspicion of a PI resistance mutation.
* Clinical condition requiring the use of a prohibited medication in association with LPV/r
* Any clinically significant disease or finding during screening that, in the investigator's opinion, would compromise participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1003 (Actual)
Dates: Start 2015-09; Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Treatment effectiveness at 48 weeks based on a composite endpoint of: i) virologic response <1000 copies/ml ii) being alive and iii) on study drug | 48 weeks
  • Treatment effectiveness at 48 weeks based on a composite endpoint of: i) virologic response <1000 copies/ml ii) being alive and iii) on study drug

SECONDARY OUTCOMES:
Treatment effectiveness based on virologic, immunologic and clinical endpoints | 96 weeks
  * Viral load suppression <1000 copies/ml (as well as <400 &<50 copies/ml where viral load can be measured on plasma) 48 weeks, 96 weeks, after treatment initiation among children under LPV/r based therapy (i.e. in completers) and at the end of the follow-up
  * Clinical failure at 48 weeks and at the end of follow-up defined as new or recurrent disease progression (WHO AIDS definition), death,
  * Immunologic failure as defined by the presence of any of the following:
    1. CD4 percentage fails to rise by 5 percentiles (or CD4 count fails to rise by at least 50 cells/mm3) during the first year of HAART.
    2. CD4 count drops by more than 50% of the peak achieved on HAART.
    3. Decline below age dependent CD4% or CD4 cells count/ml (WHO thresholds for severe immunodeficiency)
  * Retention on therapy
Rate of AEs/SAEs as measure of safety | 96 weeks
  * Rate of severe adverse events
  * Rate of AE/serious AE leading to treatment discontinuation
  * Rate of targeted AEs for lopinavir/ritonavir as well as NRTIs (examples: GI side effects, liver toxicity, ABC-associated hypersensitivity reaction, ZDV-related anaemia and neutropenia…)
Pharmacokinetics - Plasma AUC | 96 weeks
  * Plasma AUC, Tmax and C12/Cmin upon population PK modelling upon using sparse sampling
  * Exposure to LPV/r & adherence as measured by ARV levels in hair
Feasibility and acceptability questionnaires | 96 weeks
  • Questionnaire on Acceptability by caregivers and children of the new LPV based formulation , in particular taste, ease of swallowing, ease of administration, adherence
Pharmacokinetics - Tmax | 96 weeks
  * Plasma AUC, Tmax and C12/Cmin upon population PK modelling upon using sparse sampling
  * Exposure to LPV/r & adherence as measured by ARV levels in hair
Pharmacokinetics - C12/Cmin | 96 weeks
  * Plasma AUC, Tmax and C12/Cmin upon population PK modelling upon using sparse sampling
  * Exposure to LPV/r & adherence as measured by ARV levels in hair

CONTACTS AND LOCATIONS:
Overall Officials: Dalton Wamalwa, MD, Principal Investigator — University of Nairobi, P.O Box 19676 00202 Nairobi
Locations (11):
- Kenya (4):
  - AMPATH - Moi Teaching and Referral Hospital, Eldoret
  - FACES Lumumba Clinic, Kisumu
  - Gertrude's Children Hospital, Nairobi
  - Kenyatta National Hospital, Nairobi
- Tanzania (2):
  - Management and Development for Health(MDH) , at Temeke and Amana Hospitals, Dar es Salaam
  - Ifakara health Institute, Morogoro
- Uganda (5):
  - Joint Clinical research Centre, Fort Portal
  - Joint Clinical Research Centre, Gulu
  - Baylor College of Medicine, Children's Foundation - Uganda, Kampala
  - Joint Clinical research Centre, Kampala
  - Epicentre Mbarara Research Centre, Mbarara

REFERENCES:
- [Derived] Chupradit S, Wamalwa DC, Maleche-Obimbo E, Kekitiinwa AR, Mwanga-Amumpaire J, Bukusi EA, Nyandiko WM, Mbuthia JK, Swanson A; DNDi Clinical Team; Cressey TR, Punyawudho B, Musiime V; LIVING Study Team. Population Pharmacokinetics of Pediatric Lopinavir/Ritonavir Oral Pellets in Children Living with HIV in Africa. Clin Pharmacol Ther. 2024 May;115(5):1105-1113. doi: 10.1002/cpt.3174. Epub 2024 Jan 21. PMID 38247190